CLINICAL TRIAL: NCT01820715
Title: A Phase I Study of the DA-3030 Injection to Evaluate Its Safety and Explore the Efficacy for Diabetic Neuropathic Pain
Brief Title: A Study to Evaluate the Safety of DA-3030 and to Explore the Efficacy for Diabetic Neuropathic Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA3030_DN_I (Version 3.4)
Record Dates: First submitted 2013-03-15; First posted 2013-03-29 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 600㎍ of DA-3030 Injection (Experimental): 600㎍ of DA-3030 is injected once a day, for 5 continuous days.
  Interventions: Drug: 600㎍ of DA-3030 Injection
- Placebo (Placebo Comparator): Placebo(a salin drip) is injected once a day, for 5 continuous days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 600㎍ of DA-3030 Injection
  Arms: 600㎍ of DA-3030 Injection
Drug: Placebo
  Arms: Placebo

SUMMARY:
A multi-centers, placebo-controlled, randomized, double-blinded, pilot clinical trial is designed to evaluate the safety of the DA-3030 injection and to explore the efficacy for Neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* 20≤ Age ≤ 70
* Diagnosed with Type I or Type II diabetes
* HbA1c ≤ 11%
* Patients with diabetic neuropathic pain for at least 3 months
* Patients corresponding to average pain level of 4 points or mor for 24 hours evaluated with 11-point Likert scale

Exclusion Criteria:

* Neuropathic pain due to other causes
* Another stronger pain other than neuropathic pain
* Abnormality in blood pressure, weight
* Positive reaction in HIV, HBV or HCV
* A medical history of mental illness within 6 months
* The grade of BDI(Beck Depression Inventory) exceeds 21 points
* History of drug/alcohol abuse

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Abnormal score of vital signs measured by following methods: two-sample t-test, Wilcoxon rank sum test, Paired t- test, Wilcoxon signed rank test, McNemar test, Chi-squared test, or/and Fisher's exact test | 12 Weeks
Number of Subjects or Incidence with Adverse Events including Adverse Drug Event and Serious Adverse Event | 12 weeks

SECONDARY OUTCOMES:
Average pain score | 12 Weeks
  Measuring how much the subject feels pain last 24 hours on a scale of one to ten (no pain - most severe pain)
Most severe pain score | 12 weeks
  Measuring how much the subject feels pain last 24 hours on a scale of one to ten (no pain - most severe pain)
overnight pain score | 12 weeks
  Measuring how much the subject feels pain last night on a scale of one to ten (no pain - most severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Yoo Heon Ahn, M.D., Ph.D., Principal Investigator — Hanyang University; Bong Yeon Cha, M.D., Ph.D., Principal Investigator — Seoul St. Mary's Hospital, The Catholic University of Korea; Kyung Soo Ko, M.D, Ph.D., Principal Investigator — Inje University; Tae Sun Park, M.D., Ph.D., Principal Investigator — Chonbuk National University Hospital; Young Soo Park, M.D.,Ph.D., Principal Investigator — Hanyang University Guri Hospital; Choon Hee Chung, M.D., Ph.D., Principal Investigator — Wonju Christian Hospital; In Joo Kim, M.D., Ph.D., Principal Investigator — Pusan National University Hospital
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea